CLINICAL TRIAL: NCT02278809
Title: Promoting Healthy Lifestyle Behaviors in Primary Schoolchildren: Evaluation and Implementation of an Online Video Intervention for Parents
Brief Title: Promoting Healthy Lifestyle Behaviors in Schoolchildren: an Online Video Intervention for Parents
Acronym: Movie Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Flemish Agency for Care and Health (Other); Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B670201214212
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Physical Activity; Sedentary Behavior; Healthy Diet; Primary Schoolchildren; Parents; Parenting
Keywords: physical activity; screen time; vegetables; fruit; snacks; softdrink; water; fruit juice; parenting practices; online videos; intervention mapping protocol
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- waitlist control group (No Intervention): The waitlist control group parents received the online videos when the intervention period was over.
- intervention group (Experimental)
  Interventions: Behavioral: Movie Models

INTERVENTIONS:
Behavioral: Movie Models — The intervention group got acces to a private website for 4 weeks on which the online videos were placed (Week 1: fruit + water, week 2: vegetables + breakfast + supermarket, week 3: PA, week 4: SB)
  After each week, parents received a link for an online process evaluation questionnaire in which we asked how many times they watched each video, if they discussed the videos with other people, if they found them interesting, boring…
  Arms: intervention group

SUMMARY:
1. Development of a method for parents of primary schoolchildren to teach parents parenting skills to obtain health gain in the family through videos and online feedback.
2. Effect- and procesevaluation of this methodology.
3. Development of an implementation guide together with VIGEZ as primary partner and in association with partner organisations on the field.

DETAILED DESCRIPTION:
The current project aims to develop, test and implement online videos to teach effective parenting skills to parents of primary schoolchildren. This way we want to achieve health profit by stimulating PA en healthy diet, and reducing SB in children. The online videos, based on existing literature and focus group research, show parents via modeling how they can react in difficult parenting situations related to PA, SB and healthy diet. In the current study, these videos will first be tested in an effect and process evaluation study. 300 families with at least one primary schoolchild will be recruited and randomized into an intervention/control group. By using a survey at the pre-, post- and follow-up test, we will examine if parenting practices become more effective, if related parental self-efficacy enhances and if children perform more healthy behaviors after their parents watched the videos.

ELIGIBILITY:
Inclusion Criteria:

* having at least one primary schoolchild
* having a computer at home with internet access

Exclusion Criteria:

* primary schoolchild is on diet
* primary schoolchild has a physical disability which causes problems to move/sport
* being younger than 18 or older than 70
* having no internet access

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in physical activity level of children at 1 and 4 months | After 1 and 4 months
Change from Baseline in sedentary behavior of children at 1 and 4 months | After 1 and 4 months
Change from Baseline in healthy diet of children at 1 and 4 months | After 1 and 4 months

SECONDARY OUTCOMES:
Change from Baseline in performing effective parenting practices of parents at 1 and 4 months | After 1 and 4 months
Change from Baseline in parental self-efficacy concerning performing effective parenting practices at 1 and 4 months | After 1 and 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sara De Lepeleere, Ghent, Belgium

REFERENCES:
- [Derived] Van Stappen V, De Lepeleere S, Huys N, Latomme J, Verloigne M, Cardon G, Androutsos O, Manios Y, De Bourdeaudhuij I, De Craemer M. Effect of integrating a video intervention on parenting practices and related parental self-efficacy regarding health behaviours within the Feel4Diabetes-study in Belgian primary schoolchildren from vulnerable families: A cluster randomized trial. PLoS One. 2019 Dec 11;14(12):e0226131. doi: 10.1371/journal.pone.0226131. eCollection 2019. PMID 31826024
- [Derived] De Lepeleere S, De Bourdeaudhuij I, Cardon G, Verloigne M. The effect of an online video intervention 'Movie Models' on specific parenting practices and parental self-efficacy related to children's physical activity, screen-time and healthy diet: a quasi experimental study. BMC Public Health. 2017 Apr 27;17(1):366. doi: 10.1186/s12889-017-4264-1. PMID 28449658